CLINICAL TRIAL: NCT04890782
Title: Gut Microbiota in Patients With Moyamoya Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY 2021-072-01
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Moyamoya Disease; Gut Microbiota
Keywords: Moyamoya Disease; Microbiome; RNF213 p.R4810K; MRI
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MMD group: Consecutive patients diagnosed with MMD during hospitalization in Beijing Tiantan Hospital, Capital Medical University will be recruited.
- Healthy control group: Age and sex matched subjects will be invited to join the study as the control.

SUMMARY:
This study is to find out the association between gut microbiota and moyamoya disease.

DETAILED DESCRIPTION:
Moyamoya disease (MMD) is a rare cerebrovascular disorder, it is a major cause of stroke in children and young adults in Japan, Korea, and China, but its pathogenesis is not yet clear. Dysbiosis of gut microbiota may play a role in the pathological change of MMD. In this research, the investigators would perform metagenomic sequencing to find the characteristics of gut microbiota of MMD and to explore the correlations with metabolic, immune, and clinical symptoms. This research will not only help the understanding of the pathophysiology of MMD, but also may provide a reference for the selection of clinical treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MMD by DSA according to the Japanese guidelines published in 2012,
2. Stenosis or occlusion of the terminal internal carotid and the proximal middle and anterior cerebral arteries and unilateral or bilateral involvement
3. Age: 2-60 years old.

Exclusion Criteria:

1. Moyamoya syndrome,
2. Pregnancy,
3. Evidence of gastrointestinal infection/ inflammation/ obstruction
4. History of partial or total resection of small or large bowel, as well as gut reanastomosis,
5. Use of antibiotics within 2 weeks prior to symptoms onset,
6. Gastrointestinal malignancy
7. Any hospitalization within 3 months before recruitment

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Consecutive patients diagnosed with MMD during hospitalization in Beijing Tiantan Hospital will be recruited. Eligibility will be determined through a checklist of inclusion and exclusion criteria. Control group will be recruited from medical out patient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Diversity analysis of genes and species between MMD patients and the control group | Through study completion，eight months.
  Based on the gene and species composition of each sample, the Chao1 and Shannon indexes, as well as the observed OTUs (operational taxonomic units), will be calculated in order to identify the differences in gene and species diversity for each group.
Analysis of differences in intestinal microbiota between MMD patients and the control group | Through study completion，eight months.
  The Spearman correlation coefficient between genes will be calculated, and genes with strong correlation will be grouped into one cluster, as a CAG. The abundance of CAGs in each sample will be determined Furthermore, the significantly enriched species in the control and MMD groups will be enumerated for network display.
Analysis of functional differences in the intestinal microbiota of MMD patients in comparison to the control group | Through study completion，eight months.
  The LEfSe discriminant analysis will be used to screen for significant differences between groups. The dimensionality reduction will be implemented by LDA, and the impact of function difference will be evaluated to obtain the LDA score and identify significantly different functions between groups.
Analysis of metabolites of the intestinal microbiota of MMD patients in comparison to the control group | Through study completion，eight months.
  Metabolites of the intestinal microbiota between two groups

SECONDARY OUTCOMES:
Correlation analysis between gut microbiota in MMD patients and inflammatory cytokines. | Through study completion，eight months.
  IL-4,IL-10,IL-13, IFN-α, TGF-β, IL-1,IL-6, IL-17, IFN-β, IFN-γ and TNF-α
Correlation analysis between gut microbiota in MMD patients and neuroimaging markers and cognitive status. | Through study completion，eight months.
  MRI: BOLD, DWI, QSM, CUBE, ASL, T1, T2; Cognitive status: Wisdom, Attention, Memory, Linguistic fluency;
The differences of composition of gut microbiota among the genotypes (RNF213 p.R4810K) | Through study completion，eight months.
  RNF213 p.R4810K

CONTACTS AND LOCATIONS:
Overall Officials: Dong Zhang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No